CLINICAL TRIAL: NCT06334250
Title: Pulsed Field Ablation During Left Atrial Appendage Occlusion: A Randomised Controlled Trial
Acronym: PLANET-AF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision not to commence study.
Sponsor: Liverpool Heart and Chest Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRAS:327077
Record Dates: First submitted 2024-02-05; First posted 2024-03-27 (Actual); Last update posted 2024-07-19 (Actual); Status verified 2024-07

CONDITIONS: Atrial Fibrillation
Keywords: Left atrial appendage occlusion; Catheter ablation; Atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Electroporation; Left Atrial Appendage Closure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Left atrial appendage occlusion alone (Active Comparator): Left atrial appendage occlusions with the Watchman device (Boston Scientific)
  Interventions: Device: Left atrial appendage occlusion
- Combined left atrial appendage occlusion and pulsed field ablation of atrial fibrillation (Experimental): Left atrial appendage occlusion with the Watchman device (Boston Scientific) and catheter ablation of atrial fibrillation with the FaraPulse system (Boston Scientific)
  Interventions: Device: Catheter ablation of atrial fibrillation using Pulsed Field Ablation; Device: Left atrial appendage occlusion

INTERVENTIONS:
Device: Catheter ablation of atrial fibrillation using Pulsed Field Ablation — Pulsed Field Ablation of atrial fibrillation at the time of left atrial appendage occlusion
  Other Names: FaraPulse (Boston Scientific); Electroporation
  Arms: Combined left atrial appendage occlusion and pulsed field ablation of atrial fibrillation
Device: Left atrial appendage occlusion — Left atrial appendage occlusion using the Watchman device
  Other Names: Watchman device

SUMMARY:
Atrial fibrillation (AF) is the most common abnormal heart rhythm. It is also a leading cause of stroke, due to blood clots forming within an area called the 'left atrial appendage'. Usually, blood thinners (anticoagulants) are given to patients to reduce this risk. However, some patients are not able to take these medications due to a high bleeding risk. In this situation, these patients are sometimes offered a 'left atrial appendage occlusion' (LAAO) procedure - this is performed by inserting wires through the veins in the groin into the heart, then deploying a device which blocks the appendage, thus stopping blood clots from forming. There is increasing interest within our professional community of combining this procedure with another, called 'catheter ablation', which is performed to improve the symptoms of AF. This procedure uses similar access to the heart, but is not often performed in the same sitting - and often not performed at all in this patient group as they are felt to be at higher risk of complications due to bleeding or clotting. Pulsed Field Ablation (PFA) is a new technology which significantly improves safety of ablation. In this randomised controlled trial, patients referred for LAAO will be randomised to receive LAAO+PFA (intervention) or LAAO alone (control). Patients will be blinded to treatment received, which allows thorough assessment of the benefit of ablation.

DETAILED DESCRIPTION:
1. Background and Study Rationale

   Catheter ablation for atrial fibrillation (AF) has been associated with improvement in quality of life outcomes1 and even a reduction in stroke risk. Left atrial appendage occlusion (LAAO) is an effective option for preventing thromboembolic strokes in patients with AF. It is most indicated in those who have a high stroke risk but have contraindications to oral anticoagulant (OAC) therapy, such as a prior haemorrhagic stroke.

   LAAO is an invasive procedure and hence carries a degree of risk. Many of these risks are common to those encountered during a standard AF ablation procedure, which is routinely performed for symptomatic improvement (rhythm control) of AF. Both procedures require femoral venous access and trans-septal puncture to access the left atrium (LA). These procedures have traditionally been performed at separate time points, largely due to the long procedure duration for AF ablation and resulting long LA dwell time (which is associated with increased risk of thromboembolic procedural complications). However, the disadvantage is a cumulative increased risk of other complications, especially with repeated vascular access and the need for two trans-septal punctures with this approach.

   The advent of PFA as a new modality for AF ablation now means that AF ablation can be performed very quickly, with LA dwell times of 15-20 minutes compared to more conventional methods of up to 2 hours. Given that LAAO itself also requires an LA dwell time of 15-20 minutes, this makes it feasible and indeed attractive to perform both procedures simultaneously in suitable patients. Whilst this would increase the LA dwell time, it would remain comparable to prior ablation technologies (which carry a proven safety record) and would reduce the risk of other complications caused by a second procedure (e.g., vascular damage, cardiac tamponade, etc).

   The optimal patient population, and procedure-related outcomes, for this combined procedure have not been studied.
2. Hypothesis

   Combined AF ablation and LAAO results in better quality of life outcomes compared with LAAO alone.
3. Design

   Two centre, patient-blinded, randomised controlled trial
4. Inclusion and exclusion criteria

   See section below.
5. Study Methodology and Flow

   If the patient decides to participate, baseline data will be collected, and the patient will be randomised to a treatment arm. Randomisation will take place as close to the procedure as possible, however this does need to be done in advance as different equipment setups are required per arm. All patients will undergo a pre-procedural CT scan and echocardiogram, as is standard for routine clinical care - randomisation should take place AFTER the CT scan has confirmed eligibility. Following their procedure, all patients will be provided with an AliveCor monitoring device and instructed to take daily recordings, with additional recordings in the event of symptoms. These ECGs will be automatically uploaded to the KardiaPro ECG platform which the study coordinator will access to determine recurrence of arrhythmia.

   Patients will be followed up as per routine clinical care and will also have a research follow-up at 3, 6 and 12 months. At each follow-up, a discussion will take place to identify any potential study outcomes or adverse events which have occurred, and ensure the patient is not having difficulties utilising their AliveCor device. At baseline and 12 months, a quality of life questionnaire will be completed. The AliveCor device will be retrieved from the patient at 12 months.
6. Procedure Protocol

   The approach to both AF ablation and LAAO is at the discretion of the operator(s). The intent of this study is to compare outcomes with the technology itself, rather than specific techniques.

   All procedures will be performed under general anaesthesia as is routine for these cases. This allows for patient blinding - every effort must be made to ensure the patient is not informed whether or not they will be receiving ablation.

   Patients will be electrically cardioverted to sinus rhythm prior to cardiac intervention. In the intervention arm, PVI with PFA will be performed prior to LAAO. This will utilise the FaraPulse system (Boston Scientific). Typically, this involves 8 applications per pulmonary vein (4 in flower configuration and 4 in basket configuration), but additional applications may be made at operator discretion.

   LAAO will be performed in isolation in the control arm (or following PFA in the intervention arm). LAAO will be performed with the Watchman device (Boston Scientific).

   If typical atrial flutter occurs during the case, a separate RF catheter may be used to perform cavotricuspid isthmus (CTI) ablation. All other flutters will be cardioverted but not treated by ablation. In particular, the PFA catheter will not be used to attempt mitral lines or CTI ablation. 3D mapping will not be used.
7. Post Procedural ECG Monitoring

   Following their ablation and before discharge, patients will be provided with an AliveCor monitor device and will be assisted to set this up on their smartphone. This will be registered with the KardiaPro cloud to allow ECG uploading for the study. Patients will be instructed to perform a once daily 6-lead ECG, and additional ECGs in the event of symptoms suggestive of AF.
8. Outcome Measures

Primary Outcome

Change in quality of life from baseline to 12 months as measured by the AFEQT questionnaire

Secondary Outcomes

Time to AF recurrence (determined by AliveCor monitoring) Requirement for unplanned further ablation or cardioversion procedures Procedural metrics (procedure time, x-ray time, left atrial dwell time, etc) Safety outcomes - acute procedural complications, delayed procedural complications, adverse events

ELIGIBILITY:
Inclusion Criteria:

* Paroxysmal or Persistent AF, aged 18-80
* Presence of symptoms attributable to AF: EHRA 2 and above
* Clinical indication for LAAO procedure
* Own smartphone compatible with AliveCor device

Exclusion Criteria:

* Permanent AF
* Body mass index ≥40
* Previous LA ablation procedure
* Severely enlarged LA (>50mm antero-posterior diameter)
* Severely impaired left ventricular function (ejection fraction < 35%)
* Severe valvular disease
* Significant renal impairment (estimated glomerular filtration rate < 30)
* Pregnancy
* Significant frailty (Clinical Frailty Score < 5)
* Non-AF arrhythmia (e.g., atypical flutter, focal atrial tachycardia, other narrow complex tachycardias)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — All
Enrollment: 0 (Actual)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in quality of lfie | Measured at baseline and at 12 months following the procedure
  Change in quality of life from baseline to 12 months as measured by the Atrial Fibrillation Effect On Quality-Of-Life Questionnaire (AFEQT) questionnaire

SECONDARY OUTCOMES:
Time to atrial fibrillation recurrence | From the day of the procedure to end of follow-up at 12 months
  Time to atrial fibrillation recurrence, determined by AliveCor monitoring
Requirement for unplanned further ablation or cardioversion procedures | From the day of the procedure to end of follow-up at 12 months
  Requirement for unplanned further ablation or cardioversion procedures during 12 month follow-up
Procedural metrics | On the day of the left atrial appendage +/- pulsed field ablation procedure
  Procedure time, x-ray time, left atrial dwell time
Procedural safety outcomes | From the day of the procedure to end of follow-up at 12 months
  Acute procedural complications, delayed procedural complications, adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Dhiraj Gupta, MD, Principal Investigator — Liverpool Heart and Chest Hospital
Locations (1):
- Liverpool Heart and Chest Hospital, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No